CLINICAL TRIAL: NCT03186651
Title: An Open Randomized Controlled Multicenter Clinical Investigation With an Intra-vaginal Device for Stress Urinary Incontinence in Comparison to Using Standard of Care
Brief Title: An Investigation With an Intra-vaginal Device for Stress Urinary Incontinence
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Invent Medic Sweden AB (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: TVS1000
Record Dates: First submitted 2017-03-24; First posted 2017-06-14 (Actual); Last update posted 2018-04-04 (Actual); Status verified 2018-04

CONDITIONS: Stress Urinary Incontinence
Keywords: Vaginal; Medical Device; Female Stress Urinary Incontinence
MeSH Terms: conditions — Urinary Incontinence, Stress

STUDY DESIGN:
Masking Description: Open Lable
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Trans Vagina Support (Experimental): Tension Free Vaginal Support (TVS):The subjects in the TVS Group used pads during week 1 (Baseline), fitted, trained and selected device size week 2 and used the selected device size during week 3 (treatment week).
  Interventions: Device: TVS
- Standard Care (No Intervention): Standard of care (SoC): The subjects in the SoC group continued with conventional treatment i.e. using pads during week 1, 2 and 3. They were offered to use the TVS device for two weeks after completion of week 3.

INTERVENTIONS:
Device: TVS — Efficacy of a novel intra-vaginal device for temporary reduction of urine leakage in women suffering from stress urinary incontinence and to evaluate the safety and ease of use.
  Arms: Trans Vagina Support

SUMMARY:
This is a prospective, randomized, controlled, two-armed multi-center pre-market trial. Nighty-six (96) subjects will be recruited at sites in Sweden. Patients with diagnosed stress urinary incontinence (SUI), will be considered as potential study participants. After written informed consent has been acquired, a medical and surgical history, a physical examination (including pelvic examination), and a confirmation of the diagnosis of SUI will be performed, followed by a confirmation of the inclusion/exclusion criteria. The study subjects fulfilling all the eligibility criteria will thereafter be randomized 3:1 into either the TVS group or the standard of care (SoC) group.

ELIGIBILITY:
Inclusion Criteria:

1. Signed Informed Consent Form
2. Over the age of 18 years
3. Women diagnosed with stress urinary incontinence
4. Normal voiding without residual urine ≤100mL
5. Leakage of at least 10 grams per 24 hours (based on pad-weight test)
6. Provoking test with leakage

Exclusion Criteria:

1. History of dominated urgency's symptoms
2. Any contraindication for the investigational device; such as hypersensitivity to silicon rubber
3. Unexplained pelvic bleeding or vaginal discharge
4. Is hysterectomized,has a history of incontinent surgery or surgery for prolapse correction.
5. The woman is currently using prolapse ring
6. Women with prolapse reaching the hymus during coughing.
7. Pregnant or suspicion of pregnancy
8. Urinary tract or vaginal infection
9. History of not being able to use tampons
10. Neurogenic bladder dysfunction
11. The patient is to start, or change an ongoing, pelvic floor training
12. If the patient does not have a well adjusted diuretica, or is to start, or change an ongoing, diuretic treatment
13. The patient is participating in another study on SUI
14. Any other condition that as judged by the investigator may make follow-up or investigations inappropriate
15. Any patient that according to the Declaration of Helsinki is unsuitable for enrollment

Ages: 18 Years to 85 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 97 (Actual)
Dates: Start 2017-02-27 (Actual); Primary Completion 2018-02-14 (Actual); Study Completion 2018-03-28 (Actual)

PRIMARY OUTCOMES:
Absolute reduction in leakage as measured by pad weight in gram | 3 weeks
  The primary endpoint will be the absolute reduction in pad weight from the run-in week (week 1) compared with the final week (week 3). The weight of the pad is defined as the mean weight over the entire week of measurement.

SECONDARY OUTCOMES:
Success rate in % in reducing urinary leakage measured by pad weight | 3 weeks
  Overall success rate, defined as at least 70% reduction in pad weight measured in gram from run-in to the final week (week 3).
Reduction of urinary leakage episodes measured by subjective observations | 3 weeks
  Reduction of SUI episodes from the run-in week compared to the final week (week 3) by entry of subjective observations in study diary.
General impact on quality of life parameters | 3 weeks
  General impact on quality of life parameters using European Quality of Life - 5 dimensions (EQ-5D-5L) comparing week 1 and week 3.
Impact on disease specific qulity of life parameters | 3 weeks
  Disease specific Impact of Quality of life parameters, measured by the Incontinence Impact Questionnaire (IIQ-7), Urogenital Distress Inventory (UDI-6) comparing week 1 and week.

OTHER OUTCOMES:
Number of participants with treatment-related adverse events as assessed by reported events. | 3 weeks
  Possible device related adverse reactions

CONTACTS AND LOCATIONS:
Overall Officials: Aino Fianu Jonasson, MD, PhD, Principal Investigator — Kvinnokliniken Karolinska sjukhuset
Locations (4):
- Sweden (4):
  - Ladulaas Kliniska Studier, Borås
  - Kvinnokliniken Karolinska Sjukhuset, Huddinge
  - PTC-Skaraborg, Skövde
  - PTC-Göteborg, Västra Frölunda

IPD SHARING:
Plan to Share IPD: No